CLINICAL TRIAL: NCT05406622
Title: A Prospective, Multicenter, Single Blind, Randomized Controlled Trial Evaluating the Safety and Effectiveness of the MOTIV Sirolimus-Eluting Bioresorbable Vascular Scaffold Compared With Plain Balloon Angioplasty for the Treatment of Infrapopliteal Lesions
Brief Title: MOTIV BTK Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: REVA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCT6800
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MOTIV Sirolimus-Eluting Bioresorbable Scaffold (Experimental): Participants who receive the MOTIV device will be included in this arm
  Interventions: Device: MOTIV Sirolimus-Eluting Bioresorbable Scaffold
- Percutaneous Transluminal Angioplasty (PTA) (Active Comparator): Participants who receive PTA treatment will be included in this arm
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA) Device

INTERVENTIONS:
Device: MOTIV Sirolimus-Eluting Bioresorbable Scaffold — Participants will receive the MOTIV device
  Arms: MOTIV Sirolimus-Eluting Bioresorbable Scaffold
Device: Percutaneous Transluminal Angioplasty (PTA) Device — Participants will receive PTA treatment
  Arms: Percutaneous Transluminal Angioplasty (PTA)

SUMMARY:
Pre-market clinical evaluation of the MOTIV Sirolimus-Eluting Bioresorbable Scaffold for the planned treatment of infrapopliteal lesions.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria

Subjects must meet all of the following criteria to be eligible for enrollment in the trial:

1. Subject is at least 18 years of age.
2. Subject presents with symptomatic CLI classified as Rutherford category 4 or 5.
3. Subject agrees to comply with all-protocol specified procedures and follow-up assessments.
4. Subject or subject's legal representative signs an IRB/EC approved informed consent form prior to study participation.

Angiographic Inclusion Criteria

Subjects must meet the following criteria to be eligible for participation in the study:

1. Significant stenosis (>70% diameter stenosis by visual estimate) of one or two native infrapopliteal lesions; if two lesions, each lesion should be in a separate infrapopliteal vessel in the same limb. Unstented restenotic lesions are permitted.
2. Target vessel diameter between 2.5 mm and 3.75 mm and able to be treated with the available device size matrix.
3. Each target lesion is treatable by a maximum of 3 scaffolds, and all target lesions(s) combined must be treatable by a maximum of 4 scaffolds.
4. Total scaffold length among all target lesions must not exceed 120 mm (total sirolimus drug dose of 720 µg).
5. Target lesion(s) must be at least 4 cm above the ankle joint
6. Target lesion(s) are located in an area that may be stented without blocking access to patent main branches.
7. A patent inflow artery from the aorta to the target lesion free from significant stenosis (≥50% diameter stenosis by visual estimate) must be present, as confirmed by angiography.
8. Significant lesions (≥50% diameter stenosis) in inflow arteries must be treated successfully (per physician's assessment) using standard of care treatment prior to enrollment; inflow lesion treatment may be performed during the index procedure.
9. Target vessel(s) reconstitute(s) at or above the ankle or displays normal terminal branching with inline flow to at least one patent (<50% diameter stenosis by visual assessment) outflow vessel.

Exclusion Criteria:

Clinical Exclusion Criteria

Subjects will be excluded if any of the following criteria apply:

1. Subject has severe medical comorbidities or other medical, social or psychological condition that could limit subject's ability to participate in the study or is associated with a life expectancy of less than 1 year.
2. Subject has documented history of stroke within 3 months prior to the procedure.
3. Subject has history of MI, within 30 days prior to the planned index procedure.
4. Subjects with renal failure (estimated Glomerular Filtration Rate [eGFR] < 30 ml/min).
5. Subject has non-atherosclerotic disease resulting in occlusion (e.g., embolism, Buerger's disease, vasculitis).
6. Subject presents with CLI classified as Rutherford category 6.
7. Subject has acute limb ischemia, defined as symptom onset occurring less than 14 days prior to the index procedure with associated loss of sensation or motor function.
8. Subject had a major amputation that occurred less than one year prior to enrollment and subject is not independently ambulating.
9. Subject has a planned major amputation (of either leg).
10. Subject has had, or currently requires, surgical revascularization in the target vessel.
11. Subject has a planned use of adjunctive primary treatment modalities (e.g., radiation therapy, stents) in below-the-knee vessels; plaque modification technology such as the use of atherectomy, laser or cutting balloons is permitted.
12. Subject has any systemic infection or immunocompromised state.
13. Subject has a coagulation disorder, including hypercoagulability; or the subject has contraindication to anticoagulant or antiplatelet therapy.
14. Subject has a known history of heparin-induced thrombocytopenia (HIT) type II.
15. Subject has known allergy or sensitivity to scaffold or scaffold components.
16. Subject has a known allergy or sensitivity to contrast media that cannot be adequately pre-treated.
17. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
18. Subject is currently participating in another investigational drug or device clinical study that has not yet met its primary endpoint.

Angiographic Exclusion Criteria

Subjects will be excluded if any of the following criteria apply:

1. Target lesion(s) with severe calcification (PARC defined).
2. Target lesion(s) will be subjected to significant bending and axial compression.
3. Target lesion(s) located in highly tortuous vessels.
4. Target lesion(s) previously stented (in-stent restenotic lesion).
5. Target vessel(s) has any other significant lesions (≥50% diameter stenosis by visual assessment) that is not a target lesion.
6. Target vessel previously treated within 3 months prior to index procedure
7. Angiographic evidence of thromboembolism in target limb
8. Inflow-limiting arterial stenoses are unsuccessfully treated or left untreated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Composite of Limb Salvage and Primary Patency | 6 Months
  Freedom from the composite of above-the-ankle amputation, target lesion occlusion, and clinically driven target lesion revascularization (CD-TLR).
Primary Safety Endpoint: Freedom from Major Adverse Limb Events (MALE) and All-Cause Peri-Operative Death (POD) | 30 Days
  Freedom from the composite of all-cause death, above-the-ankle amputation, or major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of the index limb involving the infrapopliteal arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Ehrin Armstrong, MD, Principal Investigator — Adventist Health; Andrej Schmidt, PD Dr., Principal Investigator — University Leipzig
Locations (4):
- United States (3):
  - Adventist Health, St. Helena, California
  - UnityPoint Health Trinity Bettendorf Hospital, Bettendorf, Iowa
  - Cardiovascular Medicine PC, Davenport, Iowa
- University Leipzig, Leipzig, Germany